CLINICAL TRIAL: NCT03872661
Title: A Multicenter Phase II Trial of Neoadjuvant IBI308, Bevacizumab, Plus Pemetrexed and Carboplatin Followed by Surgery in Patients With Unresectable Stage III Non-Small Cell Lung Cancer
Brief Title: Neoadjuvant IBI308, Bevacizumab, Plus Pemetrexed and Carboplatin Followed by Surgery in Unresectable Stage III NSCLC
Acronym: NIBCUN
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Si-Yu Wang, Professor, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GASTO1048
Record Dates: First submitted 2019-02-27; First posted 2019-03-13 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-12

CONDITIONS: Lung Cancer Stage III
MeSH Terms: conditions — Lung Neoplasms | interventions — sintilimab; Bevacizumab; Pemetrexed; Carboplatin; Thoracic Surgical Procedures

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Drug and surgery (Experimental): Neoadjuvant therapy followed by surgery. Neoadjuvant therapy included four drugs. IBI308 was given 200 mg iv infusion on day 1 of each 21-day cycle for 4 cycles; bevacizumab was administered at a dose of 15 mg/kg; pemetrexed was given 500 mg/m^2 i.v. injection on day 1 of each 21-day cycle for 4 cycles; carboplatin was given dosed to an area under the serum concentration-time curve (AUC) of 5 i.v. on day 1 of each 21-day cycle for 4 cycles. Surgery will be performed at least 21 days after the last dose of neoadjuvant therapy.
  Interventions: Drug: IBI308; Drug: Bevacizumab; Drug: Pemetrexed; Drug: Carboplatin; Procedure: Thoracic surgery

INTERVENTIONS:
Drug: IBI308 — IBI308 was given 200 mg iv infusion on day 1 of each 21-day cycle for 4 cycles.
  Other Names: Sintilimab
Drug: Bevacizumab — Bevacizumab was administered at a dose of 15 mg/kg on day 1 of each 21-day cycle for 4 cycles.
  Other Names: Avastin
Drug: Pemetrexed — Pemetrexed was given 500 mg/m^2 i.v. injection on day 1 of each 21-day cycle for 4 cycles.
  Other Names: Pemetrexed disodium
Drug: Carboplatin — Carboplatin was given dosed to an area under the serum concentration-time curve (AUC) of 5 i.v. on day 1 of each 21-day cycle for 4 cycles.
  Other Names: CBP
Procedure: Thoracic surgery — Surgery will be performed at least 21 days after the last dose of neoadjuvant therapy.

SUMMARY:
The purpose of this study is to studying neoadjuvant IBI308, bevacizumab, plus pemetrexed and carboplatin followed by surgery to see how well it works in treating patients with unresectable stage III non-small cell lung cancer.

DETAILED DESCRIPTION:
Concurrent chemoradiotherapy is the recommended therapeutic approach for patients with unresectable stage III non-small cell lung cancer (NSCLC), although surgery offers the chance of cure. With combined-modality therapy with radiation therapy and chemotherapy, the prognosis of stage III NSCLC remains poor. IBI308 (sintilimab) is a recombinant humanized anti-PD-1 monoclonal antibody. This study is to studying neoadjuvant IBI308, bevacizumab, plus pemetrexed and carboplatin followed by surgery to see how well it works in treating patients with unresectable stage III non-small cell lung cancer.

ELIGIBILITY:
Inclusion Criteria:

* Target population is unresectable stage III non-small cell lung cancer.
* Written informed consent provided.
* Subjects should not have a previously detected sensitizing EGFR mutation or ALK fusion oncogene.
* Male and female patients aged ≥18 years, < 75 years.
* Able to comply with the required protocol and follow-up procedures, and able to receive oral medications.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-1.
* Life expectancy ≥12 weeks.
* Adequate hematological function: Absolute neutrophil count (ANC) ≥2.0 x 109/L, and Platelet count ≥100 x 109/L, and Hemoglobin ≥9 g/dL (may be transfused to maintain or exceed this level).
* Adequate liver function: Total bilirubin ≤ 1.5 x upper limit of normal (ULN), Aspartate aminotransferase (AST), alanine aminotransferase (ALT) ≤ 2.5 x ULN in subjects without liver metastases; ≤ 5 x ULN in subjects with liver metastases.
* Adequate renal function: Serum creatinine ≤ 1.25 x ULN, or ≥ 60 ml/min.
* Female subjects should not be pregnant or breast-feeding.

Exclusion Criteria:

* Known severe hypersensitivity to IBI308 or any of the excipients of this product.
* Prior therapy with anti-PD-1, anti-PD-L1, anti-PD-L2, or anti-CTLA-4 antibody (including any other antibody or drug specifically targeting T-cell co-stimulation or checkpoint pathways).
* Prior chemotherapy or radiotherapy.
* Subjects with active, known or suspected autoimmune disease. Subjects in conditions not expected to recur in the absence of an external trigger, or not requiring systemic treatment are permitted to enroll.
* Subjects with a condition requiring systemic treatment with either corticosteroids (>10 mg daily prednisone equivalent) or other immunosuppressive medications within 14 days of first administration of study treatment. Inhaled or topical steroids, and adrenal replacement steroid doses > 10 mg daily prednisone equivalent, are permitted in the absence of active autoimmune disease.
* Inability to comply with protocol or study procedures.
* A serious concomitant systemic disorder that, in the opinion of the investigator, would compromise the patient's ability to complete the study.
* A serious cardiac condition, such as myocardial infarction within 6 months, angina, or heart disease.
* History of another malignancy in the last 5 years with the exception of the following: other malignancies cured by surgery alone and having a continuous disease-free interval of 5 years are permitted. Cured basal cell carcinoma of the skin and cured in situ carcinoma of the uterine cervix are permitted.
* Any unstable systemic disease (including active infection, uncontrolled hypertension, unstable angina, congestive heart failure, myocardial infarction within the previous year, serious cardiac arrhythmia requiring medication, hepatic, renal, or metabolic disease).
* Patient who has active serious infection (e.g. pyrexia of or 38.0℃ over)
* Known history of testing positive for human immunodeficiency virus (HIV) or known acquired immunodeficiency syndrome (AIDS).
* Known history of active Hepatitis B or C.
* Women who are pregnant or nursing.
* Evidence of any other disease, neurological or metabolic dysfunction, physical examination or laboratory finding giving reasonable suspicion of a disease or condition that contraindicated the use of an investigational drug or puts the subject at high risk for treatment-related complications.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2019-03-01 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Resectability rate | 3 months
  Resectability rate was defined as the percentage of patients who were able to undergo surgery after induction.

SECONDARY OUTCOMES:
Number of participants with perioperative complications | 2 years
  Safety

OTHER OUTCOMES:
Event-free survival | 2 years
  Event-free survival was defined as the time from registration to disease progression (local relapse or distant metastases) or death from any cause, whichever came first.
Overall survival | 2 years
  Overall survival was assessed from randomization to death as a result of any cause.

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China